CLINICAL TRIAL: NCT07112625
Title: Impact of Therapeutic Education for Type 2 Diabetic Patients During Ramadan. : A Randomized Controlled Trial
Brief Title: Impact of Therapeutic Education for Type 2 Diabetic Patients During Ramadan.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Imen Zemni, Medical Doctor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMONASTIR2
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- education and coaching (Active Comparator): education before ramadan fasting and during ramadan
  Interventions: Other: education and coaching
- education only (Active Comparator): education before ramadan fasting only
  Interventions: Other: education
- Controle (No Intervention): No intervention

INTERVENTIONS:
Other: education and coaching — education associated to coaching
  Arms: education and coaching
Other: education — education without coaching
  Arms: education only

SUMMARY:
This randomized controlled trial evaluates the impact of therapeutic education, with or without personalized coaching, on clinical and biological outcomes in patients with type 2 diabetes during Ramadan fasting. Participants were randomly assigned to three groups: Control (usual care), Education Only, and Education plus Coaching. All received a 30-minute pre-Ramadan education session; the Education plus Coaching group also had follow-up telephone consultations. Outcomes included HbA1c, fasting blood glucose, cholesterol, BMI, and blood pressure measured before and after Ramadan. The study aims to assess whether structured education and ongoing coaching help patients fast safely and maintain better metabolic control.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetic patients taking oral treatment who intended to fast during Ramadan and agreed to participate in the study.

Exclusion Criteria:

* Patients with severe comorbidities (renal failure, recent coronary disease, cognitive impairement) and those classified as very high risk for fasting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
HbA1c Level after ramadan | From enrollment (two weeks before ramadan219) to two weeks after ramadan 2019
  the level of HbA1c after ramadan
HbA1c level after ramadan | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Medical Doctor, Study Chair — Fattouma bourguiba university hospital of Monastir
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No